CLINICAL TRIAL: NCT00810628
Title: Depression in Parkinson's Disease: A Pilot Project Using Cognitive Behavioral Therapy (CBT) to Improve Depression and Coping
Brief Title: Cognitive Behavioral Therapy for Depression in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: Julie Carter, MS, ANP, Oregon Health & Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OHSUIRB4613
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2008-12

CONDITIONS: Parkinson's Disease; Depression
Keywords: Parkinson's disease; depression; Parkinson's disease with mild to moderate depression.
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects in same investigative group with same CBT intervention.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Individual interviews and group discussion/training.

SUMMARY:
The purpose of this pilot program is to develop and evaluate a new treatment program for depression in Parkinson's disease (PD). The treatment uses Cognitive Behavior Therapy(CBT)to teach patients how to become more aware of their thoughts and feelings and to change thinking patterns and behaviors that may be related to depressive symptoms. This is the first time that this treatment has been used in a group setting for depression in PD.

Target population is patients in the Movement Disorders Clinic at Oregon Health & Science University who have Parkinson's disease and mild to moderate depression.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, mild to moderate depression, seen at Oregon Health & Science University

Exclusion Criteria:

* Suicidal
* Cognitive impairment with MOCA <26

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The change in CESD score | Baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie H. Carter, MS, Principal Investigator — Oregon Health and Science University; Kristine Hanna, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Dobkin RD, Allen LA, Menza M. Cognitive-behavioral therapy for depression in Parkinson's disease: a pilot study. Mov Disord. 2007 May 15;22(7):946-52. doi: 10.1002/mds.21455. PMID 17377926